CLINICAL TRIAL: NCT01602367
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 2B Trial to Evaluate the Safety and Efficacy of BMS-823778 in Overweight and Obese Subjects With Inadequately Controlled Hypertension
Brief Title: Safety and Efficacy Study of BMS-823778 to Treat Uncontrolled High Blood Pressure in Overweight and Obese Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB121-008; 2012-000509-54 (EudraCT Number)
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — BMS-823778

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: BMS-823778 (2mg) (Experimental)
  Interventions: Drug: BMS-823778
- Arm2: BMS-823778 (6mg) (Experimental)
  Interventions: Drug: BMS-823778
- Arm 3: BMS-823778 (15mg) (Experimental)
  Interventions: Drug: BMS-823778
- Arm4: Placebo (Experimental)
  Interventions: Drug: Placebo matching with BMS-823778

INTERVENTIONS:
Drug: BMS-823778 — Capsules, Oral, 2 mg, Once daily, 12 weeks
  Arms: Arm 1: BMS-823778 (2mg)
Drug: BMS-823778 — Capsules, Oral, 6 mg, Once daily, 12 weeks
  Arms: Arm2: BMS-823778 (6mg)
Drug: BMS-823778 — Capsules, Oral, 15 mg, Once daily, 12 weeks
  Arms: Arm 3: BMS-823778 (15mg)
Drug: Placebo matching with BMS-823778 — Capsules, Oral, 0 mg, Once daily, 12 weeks
  Arms: Arm4: Placebo

SUMMARY:
The purpose of this study is to determine whether BMS-823778 is safe and effective in the treatment of hypertension in overweight and obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Qualifying seated blood pressure between ≥90 and ≤105 mmHg diastolic AND ≤155 mmHg systolic
* Mean 24-hour diastolic blood pressure ≥85 mmHg
* Body mass index (BMI) ≥27 kg/m2
* If receiving an oral anti-hyperglycemic medication or a cholesterol lowering medication, receiving a stable dose for at least 6 weeks

Exclusion Criteria:

* History of Cushing's disease or syndrome, or Addison's disease
* Glycosylated hemoglobin (HbA1c) ≥10%
* Cerebrovascular insult, unstable angina, or myocardial infarction (MI) within 6 months
* History of impaired renal or hepatic function
* BMI ≥50 kg/m2
* Any injectable antihyperglycemic agent (such as insulin) within 16 weeks
* Currently receiving more than one class of antihypertensive agents within 4 weeks
* Daily use of nonsteroidal anti-inflammatory agents within 1 week
* Use of androgen medications, including topical preparations, within 6 weeks
* Diagnosis or history of breast cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The dose-dependent trend among doses of BMS-823778 and placebo by assessing the change from baseline in 24-hour ambulatory diastolic blood pressure following 12 weeks of double-blind treatment | At Day -7 (baseline) and Week 12

SECONDARY OUTCOMES:
Change in 24-hour ambulatory systolic blood pressure (SBP)(evaluation of the dose-dependent trend) | At Day -7 (baseline) and Week 12
Change in 24-hour ambulatory diastolic blood pressure (DBP) | At Day -7 (baseline) and Week 12
Change in 24-hour ambulatory SBP | At Day -7 (baseline) and Week 12
Change in ambulatory daytime and nighttime DBP | At Day -7 (baseline) and Week 12
Change in ambulatory daytime and nighttime SBP | At Day -7 (baseline) and Week 12
Change in seated DBP | At Day -7 (baseline) and Week 12
Change in seated SBP | At Day -7 (baseline) and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (32):
- United States (21):
  - Nea Baptist Clinic, Jonesboro, Arkansas
  - Local Institution, Los Angeles, California
  - Desert Medical Group Inc., Palm Springs, California
  - Local Institution, Coral Gables, Florida
  - Local Institution, Atlanta, Georgia
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Local Institution, New Orleans, Louisiana
  - Anderson And Collins Clinical Research, Inc., Edison, New Jersey
  - Premier Research, Trenton, New Jersey
  - Syracuse Preventive Cardiology, Syracuse, New York
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Pharmquest, Llc, Greensboro, North Carolina
  - Pmg Research Of Salisbury, Salisbury, North Carolina
  - Local Institution, Shelby, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Sterling Research Grp, Ltd., Cincinnati, Ohio
  - Local Institution, Greenville, South Carolina
  - Local Institution, Layton, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
- Colombia (5):
  - Local Institution, Barranquilla
  - Local Institution, Bucaramanga
  - Local Institution, Cartagena
  - Local Institution, Manizales
  - Local Institution, Medellín
- Hungary (3):
  - Local Institution, Balatonfüred
  - Local Institution, Budapest
  - Local Institution, Debrecen
- Local Institution, Ponce, Puerto Rico
- Sweden (2):
  - Local Institution, Ödeshög
  - Local Institution, Stockholm

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx